CLINICAL TRIAL: NCT03981003
Title: Serum Neurofilament-light Chain and Glial Fibrillary Acidic Proten (GFAP) Levels in Patients From the OFSEP Cohort at Different Landmarks of Multiple Sclerosis
Brief Title: Serum Neurofilament-light Chain and GFAP Levels in Patients From the OFSEP Cohort at Different Landmarks of Multiple Sclerosis
Acronym: NeurofilMS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CIVI/2018/ET-02
Record Dates: First submitted 2019-05-23; First posted 2019-06-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Neurofilament-light chain; Glial fibrillary Acidic Protein (GFAP)
MeSH Terms: conditions — Multiple Sclerosis; Charcot-Marie-Tooth disease, Type 1F | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS Patients
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — 2 x 4 ml tubes blood to screen for serum Neurofilament Light Chain and GFAP levels

SUMMARY:
The investigators hypothesize that serum neurofilament-light chain (NfL) levels can provide information about the level of activity and progression of Multiple Sclerosis at different stages and landmarks of the disease.

In addition, Glial Fibrillary Acidic Protein (GFAP) has also been identified as another serum biomarker of disability in MS.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed.
* The patient must have given their informed and signed consent.
* The patient must be insured or beneficiary of a health insurance plan.
* The patient is at least (≥)15 years old.
* The patient has MS according to diagnosis criteria (Thompson et al. 2017) and:

  * Participates to the OFSEP-HD cohort (ancillary study);
  * Has a Expanded Disability Status Scale score comprised between 0 - 7.0;
  * With or without Disease Modifying Drug;
  * For Work Package 3: patients enrolled in any OFSEP-HD centre that meet landmark criteria for an active MS (relapse, or Expanded Disability Status Scale progression, or active MRI) during follow-up;
  * For Work Package 4: patients with a stable disease enrolled in OFSEP-HD study in Nîmes or Nantes University Hospitals.

Exclusion Criteria:

* Within the past three months, the patient has participated in another interventional study that may interfere with the results or conclusions of this study.
* The patient is in an exclusion period determined by a previous study.
* The patient is under judicial protection.
* The patient refuses to sign the consent.
* It is impossible to correctly inform the patient (inability to understand the study, language problem).
* The patient is pregnant or breast-feeding.
* The patient is under 15 years old.
* Inability to answer questionnaires.
* Clinically isolated syndrome (CIS) that does not meet the criteria of MS.
* Radiologically isolated syndrome (RIS).
* Patient with Neuromyelitis optica spectrum disorder.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of consecutive patients over 15 years of age, of both sexes, recruited during consultations for a CIS, RRMS or progressive MS at the Neurology department of 30 OFSEP centres and of Nîmes and Nantes University Hospitals. The patients recruited will have an EDSS score comprised between 0 - 7.0.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Serum Neurofilament Light Chain level in patients with evolving disease compared to those with stable disease | Inclusion
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with evolving disease compared to those with stable disease | 6 months
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with evolving disease compared to those with stable disease | 12 months
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 12 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with evolving disease compared to those with stable disease | 18 months
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with evolving disease compared to those with stable disease | 2 years
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 3 years
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 4 years
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 5 years
  pg/mL; measured by digital ELISA
GFAP level in patients with evolving disease compared to those with stable disease | 6 years
  pg/mL; measured by digital ELISA

SECONDARY OUTCOMES:
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | Inclusion
  pg/mL; measured by digital ELISA
GFAP level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 6 months
  pg/mL; measured by digital ELISA
GFAP level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 3 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 4 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 5 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 6 year
  pg/mL; measured by digital ELISA
GFAP level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 18 months
  pg/mL; measured by digital ELISA
GFAP level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 2 years
  pg/mL; measured by digital ELISA
GFAP level in patients with disease activity (relapse or MRI activity determined by the presence of at least one T1 Gad+ lesion or at least one new T2 lesion ≤ 3 months) compared to stable patients. | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
GFAP level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
GFAP level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
GFAP level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
GFAP level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with progressive disease measured by Expanded Disability Status Scale (1 point until 5.5 and 0.5 point after 5.5) compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
GFAP level in patients with relapse compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapse compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
GFAP level in patients with relapse compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapse compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
GFAP level in patients with relapse compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapse compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
GFAP level in patients with relapse compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapse compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
GFAP level in patients with relapse compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
GFAP level in patients with isolated MRI activity compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
GFAP level in patients with isolated MRI activity compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 2 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement compared to stable patients | 2 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement compared to stable patients | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with stable disease (no evidence of disease activity (NEDA) and no evidence of disease progression (NEP) from 200 patients from the OFSEP-HD cohort | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in progressive MS patients with no evidence of disease progression (NEP) from the OFSEP-HD cohort with stable disease | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease evolution (relapse, disability progression or MRI activity) | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease evolution (relapse, disability progression or MRI activity) | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease evolution (relapse, disability progression or MRI activity) | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease evolution (relapse, disability progression or MRI activity) | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease evolution (relapse, disability progression or MRI activity) | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease evolution (relapse, disability progression or MRI activity) | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease evolution (relapse, disability progression or MRI activity) | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease evolution (relapse, disability progression or MRI activity) | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease evolution (relapse, disability progression or MRI activity) | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease evolution (relapse, disability progression or MRI activity) | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity) | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease activity (relapse or MRI activity) | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse, or MRI activity) | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease activity (relapse, or MRI activity) | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity) | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease activity (relapse or MRI activity) | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity) | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease activity (relapse or MRI activity) | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with disease activity (relapse or MRI activity) | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with disease activity (relapse or MRI activity) | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapses | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with relapses | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapses | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with relapses | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapses | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with relapses | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapses | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with relapses | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with relapses | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with relapses | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with MRI activity | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with MRI activity | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with MRI activity | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with MRI activity | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with MRI activity | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with MRI activity | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with MRI activity | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with MRI activity | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with MRI activity | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with MRI activity | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity and Gadolinium-enhancement | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity and Gadolinium-enhancement | 2 years
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement | 6 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement | 6 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement | 1 year
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement | 1 year
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement | 18 months
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement | 18 months
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain level in patients with isolated MRI activity without Gadolinium-enhancement | 2 years
  pg/mL; measured by digital ELISA
Serum GFAP level in patients with isolated MRI activity without Gadolinium-enhancement | 2 years
  pg/mL; measured by digital ELISA
Level of disability | Inclusion
  Expanded Disability Status Scale (EDSS); scale 1= no disability to 10 = death from multiple sclerosis
Level of disability | Relapse (measured up to 2 years)
  Expanded Disability Status Scale (EDSS); scale 1= no disability to 10 = death from multiple sclerosis
Severity of multiple sclerosis | EDSS progression (measured up to 2 years)
  Multiple Sclerosis Functional Composite
Severity of multiple sclerosis | Active MRI (measured up to 2 years)
  Multiple Sclerosis Functional Composite
Generic health status | Inclusion
  EuroQol 5 dimension questionnaire (EQ-5D)
Generic health status | Relapse (measured up to 2 years)
  EuroQol 5 dimension questionnaire (EQ-5D)
Generic health status | EDSS progression (measured up to 2 years)
  EuroQol 5 dimension questionnaire (EQ-5D)
Generic health status | active MRI (measured up to 2 years)
  EuroQol 5 dimension questionnaire (EQ-5D)
Use of Disease Modifying Drugs | Inclusion
  Categorized by class type of treatment (1st line, 2nd line and 3rd line therapies)
Use of Disease Modifying Drugs | 6 monrths
  Categorized by class type of treatment (1st line, 2nd line and 3rd line therapies)
Use of Disease Modifying Drugs | 1 year
  Categorized by class type of treatment (1st line, 2nd line and 3rd line therapies)
Use of Disease Modifying Drugs | 18 months
  Categorized by class type of treatment (1st line, 2nd line and 3rd line therapies)
Use of Disease Modifying Drugs | 2 years
  Categorized by class type of treatment (1st line, 2nd line and 3rd line therapies)
Serum Neurofilament Light Chain in 800 patients from the OFSEP cohort including Multiple Sclerosis patients at different stages and Neuromyelitis optica spectrum disorder patients | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP in 800 patients from the OFSEP cohort including Multiple Sclerosis patients at different stages and Neuromyelitis optica spectrum disorder patients | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain in 800 patients from the OFSEP cohort including Multiple Sclerosis patients at different stages and Neuromyelitis optica spectrum disorder patients | Month 6
  pg/mL; measured by digital ELISA
Serum GFAP in 800 patients from the OFSEP cohort including Multiple Sclerosis patients at different stages and Neuromyelitis optica spectrum disorder patients | Month 6
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain in 400 patients from the OFSEP cohort with a Clinically Isolated Syndrome at inclusion | Inclusion
  pg/mL; measured by digital ELISA
Serum GFAP in 400 patients from the OFSEP cohort with a Clinically Isolated Syndrome at inclusion | Inclusion
  pg/mL; measured by digital ELISA
Serum Neurofilament Light Chain in 400 patients from the OFSEP cohort with a Clinically Isolated Syndrome at inclusion | Month 6
  pg/mL; measured by digital ELISA
Serum GFAP in 400 patients from the OFSEP cohort with a Clinically Isolated Syndrome at inclusion | Month 6
  pg/mL; measured by digital ELISA
Create biobank | Inclusion
  Blood samples
Create biobank | 6 months
  Blood samples
Create biobank | 1 year
  Blood samples
Create biobank | 18 months
  Blood samples
Create biobank | 2 years
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU Nimes
Locations (28):
- France (27):
  - CHU d'Amiens, Amiens
  - CHU de Besancon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Lyon, Lyon
  - Hopital Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - CHU de Nimes, Nîmes
  - Fondation Rothschild, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Saint Antoine, Paris
  - CH de Poissy, Poissy
  - CHU de Potiers, Potiers
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No